CLINICAL TRIAL: NCT06872515
Title: Impact of Prehabilitation in Oncology Via Exercise- Esophageal
Brief Title: Impact of Prehabilitation in Oncology Via Exercise- Esophageal (IMPROVE-Esophageal)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Melanie Potiaumpai, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY24120028
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer; Esophageal Carcinoma
Keywords: Prehabilitation; Exercise; Esophageal cancer; Neoadjuvant chemotherapy; Pre-surgical exercise
MeSH Terms: conditions — Esophageal Neoplasms; Motor Activity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based prehabilitation exercise and nutrition (PRE) (Experimental): Interventions will include:
  * Up to 8 weeks of 3-5 times per week resistance training and 3-5 times per week of aerobic training.
  * Ensure Complete nutrition supplement drinks: 2 per day starting on the same day the exercise begins, up until 5 days prior to surgery.
  Interventions: Behavioral: Exercise and Nutrition
- Usual Care (CONT) (Active Comparator): The CONT group will not receive any intervention during study participation and undergo usual medical treatment and surveillance during the duration of the study.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Exercise and Nutrition — The exercise and nutrition intervention will last up to 8 weeks and will include:
  * 3-5 times per week of resistance training and 3-5 times per week of aerobic training. The prescribed exercise will be personalized based on the participant's baseline functionality.
  * Ensure Complete nutrition supplement drinks: 2 per day starting on the same day the exercise begins, up until 5 days prior to surgery.
  Arms: Home-based prehabilitation exercise and nutrition (PRE)
Behavioral: Usual Care Group — The CONT group will not receive any intervention during study participation and undergo usual medical treatment and surveillance during the duration of the study.
  Arms: Usual Care (CONT)

SUMMARY:
The goal of this study is to determine the feasibility of a prehabilitation exercise and nutrition program (exercise and nutrition before a medical treatment) in adults with esophageal cancer before surgery (esophagectomy). The pre-surgery exercise and nutrition program will include resistance and aerobic training and nutrition supplementation during the weeks before surgery. We will also assess pre-surgical care needs in adults with esophageal cancer. Researchers will compare the exercise and nutrition intervention to usual care- which is standard medical care and post-surgery surveillance/follow-up to understand the impact of exercise and nutrition before surgery. We will follow-up with participants before surgery, and after surgery at 2 weeks, 6 weeks, and 4-months at appointments that coincide with clinical follow-ups.

The main questions of this trials are:

* Is exercise and nutrition supplementation before surgery for esophageal cancer feasible and acceptable to patients?
* How does exercise and nutrition supplementation before surgery change physical function and psychosocial health?
* What are important pre-surgical needs for adults with esophageal cancer?

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥ 18 years old
* Diagnosed with esophageal cancer
* Identified as esophagectomy surgery candidates at Hillman Cancer Center or UPMC Shadyside
* ≥ 2 weeks until scheduled esophagectomy
* ECOG Performance Status Scale score of ≤ 2
* Ability to provide written informed consent
* Ability to understand, speak, and read English.

Exclusion Criteria:

* Evidence in the medical record of an absolute contraindication for exercise (e.g., Heart insufficiency > NYHA III or uncertain arrhythmia; uncontrolled hypertension; reduced standing or walking ability)
* Any other comorbidities or musculoskeletal complications that preclude participation in the exercise programs as deemed by the exercise interventionist
* Receiving non-esophagectomy related chemotherapy and/or radiotherapy
* Active infections, hemorrhages, and cytopenias that could place surgical patients at risk for further adverse events, deemed by the exercise interventionist, physician, and/or nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention | From enrollment through surgical admission, up to 8 weeks
  Acceptability is defined as the proportion of approached participants who agree to participate and complete the baseline assessments and be randomized.
Adherence to Intervention | From enrollment through surgical admission, up to 8 weeks
  Exercise adherence will be calculated as the proportion of completed exercise sessions over the number of prescribed sessions.
Feasibility of Intervention | From enrollment through surgical admission, up to 8 weeks
  The intervention will be considered feasible if 50% of participants complete approximately 70% of prescribed prehabilitation sessions prior to their surgical admission.

SECONDARY OUTCOMES:
Six-minute walk test (6MWT) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Cardiorespiratory fitness will be measured using the six minute walk test. The 6MWT is an objective evaluation of functional exercise capacity. Its results are highly correlated with those of the 12-minute walk test from which it was derived and with those of cycle ergometer or treadmill-based exercise tests.
2-Minute Step Test | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Cardiorespiratory fitness will be measured with the 2-minute step test. Participants will be marching in place for 2 minutes and are encouraged to use a chair for balance or do the assessment seated if standing is too difficult. They should be lifting their legs about 6 inches off the ground, as if they were stepping onto a curb from the road. The tester will count the number of times the participant raises their right leg off the ground.
30-second chair stand test (30CST) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Lower body strength will be evaluated using the 30 second chair stand test. The participant is seated in the middle of the chair, back straight, feet approximately shoulder width apart and placed on the floor. Arms are crossed at the wrists and held against the chest. At the signal "go," the participant rises to a full body stand and then returns to the initial seated position. The participant is encouraged to complete as many full stands as possible within 30 seconds.
Timed-Up-and-Go (TUG) test | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The TUG evaluates lower body strength, balance, and agility. The patient sits in a chair and on the command "go", the patient rises from the chair, walks 3 meters at a self-selected pace, turns around an obstacle, walks back to the chair and sits down. Test results may also be quantified assessing the time (seconds) needed to complete the assessment.
Frail Scale | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The FRAIL Scale is a short, five item assessment designed to identify frailty without face-to-face administration. The questions address Fatigue, Resistance, Ambulation, Illness, and Loss of weight (FRAIL). Scores range from 0 (robust heath status) to 5 (frail) with an intermediate category for pre-frail. Research has shown that within the geriatric fracture population, higher scores on this assessment have been shown to be associated with increased length of hospitalization, surgical complications, and more likely discharge to a rehabilitation facility rather than home making it a helpful short screen to gauge risk in the surgical population.
Handgrip assessment | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Maximum capacity to squeeze with each hand may be assessed using a hand grip dynamometer. Each hand may be assessed three times.
Short Physical Performance Battery (SPPB) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The SPPB is a short battery of performance tests of lower extremity functioning. The tests measure gait speed, standing balance, and lower extremity strength and power. To test gait speed, patients are instructed to walk an 8-foot walking course at their usual pace with assistive devices if needed. Four progressively more challenging positions are used to test balance (bipedal [feet next to each other], semi-tandem [one foot slightly in front of the other], and full tandem [one foot in front of the other]). To test lower extremity strength, patients are asked to stand up and sit down five times as quickly as possible and are timed from the initial sitting position to the final standing position at the end of the fifth stand.
Actigraph accelerometry | Baseline, 2 Weeks post esophagectomy, and 4 Months post esophagectomy
  Physical activity may be measured objectively using wearable accelerometry. Accelerometer data will include estimated average metabolic equivalents expended daily and in hours/week as well as time in sedentary, low, moderate, and vigorous activity.
SARC-F Sarcopenia scale | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The SARC-F questionnaire is a short 5-item battery containing observational assessments that is a rapid diagnostic test for sarcopenia. There are 5 SARC-F components: Strength, Assistance with walking, Rise from a chair, Climb Stairs, and Falls.
  Min = 0; Max = 10; higher score = higher risk for sarcopenia
Carbon Monoxide (CO) assessment | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Expired carbon monoxide will be evaluated using a CO analyzer (coVita Smokerlyzer Breath CO Test). The CO assessment is a rapid and noninvasive method quantify CO in the blood and illustrate current smoking habits.
Edmonton Frail Scale (EDS) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The Edmonton Frail Scale is a reliable measure for frailty that is easy to use, captures the multidimensional aspects of fatigue, and presents the level of frailty along a continuum so that change over time can be captured. The semi-structured interview collects data across 9 frailty domains: cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance. Scores fall within one of 5 categories (not frail, vulnerable, mild frailty, moderate frailty, severe frailty) and range from 0 (not frail) to 17 (severe frailty).
Demographics | Baseline
  Demographics may be collected at baseline via self-reported survey. These include date of birth, education, income, zip code, and household composition.
Injury History Survey (EX Cohort only) | Time of Admission
  Developed to assess injuries as well as discomfort from exercise. This survey will be administered to the EX cohort at the end of the intervention period at timepoint T1.
EORTC QLQ-C30 Quality of Life (QoL) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  QoL may be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It includes five multi- item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties. Scores are derived according to the EORTC scoring manual.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Multidimensional Fatigue Inventory | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Fatigue may be assessed with the Multidimensional Fatigue Inventory (MFI) which is a 20-item, multidimensional self-assessment questionnaire. It covers five different dimensions of fatigue (general, physical, reduced activity, reduced motivation, and mental). Scores are derived by summing the answers (five-stage scale) of the appropriate items.
  Min = 20; Max = 100; higher score = less fatigue
Godin Leisure Time Exercise | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Physical activity patterns during a patient's leisure time may be assessed using the Godin Leisure Time Exercise questionnaire. The questionnaire asks patients to recall, during a seven-day period, the frequency to which they participated in strenuous, moderate, and mild exercise. The Godin questionnaire is short and easy to complete.
  Min = 0; Max = none; higher score = more activity
PROMIS Smoking Assessment | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Smoking history and habits may be assessed using the PROMIS smoking assessment questionnaires. The questionnaire asks patients about their smoking habits, quit attempts, health expectations, and coping expectations.
PROMIS Cognitive Function- Short Form | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  Cognitive function may be measured by the 8-item PROMIS questionnaire. The questionnaire assesses patient-perceived cognitive deficits including mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions.
  Min = 8; Max = 40; higher score = better cognitive function
PG-SGA Nutrition Assessment- Short Form | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The Patient-Generated Subjective Global Assessment (PG-SGA) is a patient-reported instrument for assessment of nutrition status in patients with cancer. The PG-SGA short form is completed by patients and screens for nutritional risk and deficit.
  Min = 0, Max = 36; higher score = worse nutrition status
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in patients on cancer clinical trials. The PRO-CTCAE item library contains 124 items representing 78 symptomatic toxicities. Specific items can be selected to create an individualized form specific to a disease or treatment group.
Healthcare utilization | Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  To assess the impact of NAT and esophagectomy on healthcare utilization, participants may complete a validated healthcare utilization form.
Pre-Treatment Resources Assessment | Baseline
  This assessment may collect information on participants' knowledge of available supportive care resources prior to treatment and information they receive from their healthcare providers.
Brief Pain Inventory (BPI) | Baseline, Time of Admission, and 2 Weeks/6 Weeks/4 Months post esophagectomy
  The BPI is a 9-item, self-assessment questionnaire that has been largely validated. The BPI measures both the intensity of pain (sensory dimension) and interference of pain in the participant's life (reactive dimension). It also asks the participant about pain relief, pain quality, and participant perception of the cause of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Potiaumpai, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No